CLINICAL TRIAL: NCT04048824
Title: Inhibitory Learning vs. Habituation: Models of Exposure Therapy
Brief Title: Optimizing Exposure Therapy for Anxiety Disorders
Acronym: OptEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Optimizing Exposure
Record Dates: First submitted 2018-11-26; First posted 2019-08-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Social Anxiety Disorder; Panic Disorder
Keywords: inhibitory learning; exposure; anxiety; habituation; social anxiety; panic
MeSH Terms: conditions — Phobia, Social; Panic Disorder; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitory Learning-Based Exposure (Experimental): Participants will receive exposure therapy aimed at increasing inhibitory learning.
  Interventions: Behavioral: Inhibitory Learning-Based Exposure
- Habituation-Based Exposure (Active Comparator): Participants will receive exposure therapy aimed at reducing fear responding.
  Interventions: Behavioral: Habituation-Based Exposure

INTERVENTIONS:
Behavioral: Inhibitory Learning-Based Exposure — 9 weekly treatment sessions conducted individually with a therapist. Exposure is focused on maximizing the mismatch between participant's feared outcome and what actually occurred (i.e., expectancy violation). This condition includes techniques that incorporate associative learning principles such as exposure to multiple feared stimuli (i.e., deepened extinction), exposure variability in contexts and stimuli, occasional reinforcement, and mental reinstatement of inhibitory learning.
  Arms: Inhibitory Learning-Based Exposure
Behavioral: Habituation-Based Exposure — 9 weekly treatment sessions conducted individually with a therapist. Exposure is focused on fear reduction from initial fear ratings. This condition includes theoretically-consistent techniques such as staying in the situation until fear declines, repetition of exposures until fear has declined, and a gradual approach to feared stimuli using an exposure hierarchy.
  Arms: Habituation-Based Exposure

SUMMARY:
The study will compare the effects that two different approaches of exposure therapy have on reducing fear and anxiety in individuals with social anxiety disorder or panic disorder.

DETAILED DESCRIPTION:
A substantial number of individuals fail to achieve clinically significant symptom relief from exposure-based therapies or experience a return of fear following exposure therapy completion. The prevailing model of exposure therapy for phobias and anxiety disorders purports that fear reduction throughout exposure therapy (i.e., habituation) is reflective of learning and critical to overall therapeutic outcome. However, the amount by which fear - indexed by both self-report, behavioral, and biological correlates of fear expression - reduces by the end of an exposure trial or series of exposure trials is not a reliable predictor of the fear level expressed at follow-up assessment.

Developments in the theory and science of fear extinction, and learning and memory, indicate that 'performance during training' is not commensurate with learning at the process level. Inconsistent findings regarding fear reduction are paralleled by findings based in associative learning laboratory paradigms with animals and human samples, specifically that outward expression of fear on the one hand, and conditional associations indicative of underlying learning on the other hand, may not always change in concordance. Rather, 'inhibitory learning' is recognized as being central to extinction, rather than fear during extinction training.

The current proposal will compare the habituation-based model of exposure therapy to the competing inhibitory model of exposure that emphasizes learning theory principles.

The current study plans to recruit participants for a treatment trial consisting of two psychotherapies: (a) habituation-based exposure therapy and (b) inhibitory learning-based exposure therapy. The primary goal of this study is to determine if one theoretical approach to exposure outperforms the other in reducing symptoms.

This study is conducted with individuals meeting diagnostic criteria for social anxiety disorder or panic disorder. Participants will be randomized to either treatment condition and receive 9 sessions of individual psychotherapy focused on either of these disorders. If individual meets diagnostic criteria for both disorders, treatment will be focused on the primary presenting disorder. Participants will complete four assessments over the course of the study, at pre-treatment, mid-treatment, post-treatment, and three-month follow-up. Pre-treatment, mid-treatment, and post-treatment assessments occur over two days, while three-month follow-up requires only a single day and is conducted remotely.

These assessments will include semi-structured interviews, self-report questionnaires, and laboratory paradigms designed to examine fear learning processes.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking treatment for social anxiety or panic disorder and demonstration of elevated scores using standardized self-report measures and diagnostic interview
2. Age 18 to 65
3. Either stabilized on psychotropic medications or medication-free
4. English-speaking
5. Access to telehealth resources (for Zoom treatment sessions after March 2020 due to COVID-19)

Exclusion criteria include:

1. Patient report of serious medical conditions - such as respiratory (e.g., chronic obstructive pulmonary disease), cardiovascular, pulmonary, neurological, muscular-skeletal diseases - or pregnancy
2. Active suicidal ideation or self-harm in the past year; history of suicide attempts in the last 10 years
3. History of bipolar disorder, psychosis, mental retardation or organic brain damage
4. Substance abuse/dependence within last 6 months
5. Concurrent therapy focused on anxiety. Participants are allowed to be in other forms of therapy, provided the therapy does not focus on anxiety (e.g., supportive counseling) and they have been stabilized on this alternative therapy for at least 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in clinician-rated severity of social anxiety or panic disorder | Pre-treatment to post-treatment (10 weeks), to follow-up (24 weeks)
  Clinician severity rating (0-8) of social anxiety or panic disorder using the Structured Clinical Interview for DSM-5 (SCID-5).
Change in self-reported symptom severity of social anxiety or panic disorder | Pre-treatment to post-treatment (10 weeks), to follow-up (24 weeks)
  Self-reported symptom severity of social anxiety disorder using the Liebowitz Social Anxiety Scale (LSAS) or panic disorder using the Panic Disorder Severity Scale-Self Report (PDSS-SR).

SECONDARY OUTCOMES:
Change in fear extinction generalization as measured by expectancy of unconditional stimuli during conditional stimuli presentation. | Pre-treatment to post-treatment (9 weeks)
  Change in responsiveness to fear generalized from various, perceptually similar stimuli collected during a laboratory fear paradigm.
Change in fear extinction generalization as measured by skin conductance. | Pre-treatment to post-treatment (9 weeks)
  Change in skin conductance to fear generalized from various, perceptually similar stimuli collected during a laboratory fear paradigm. (Discontinued March 2020 due to COVID-19)
Change in fear extinction generalization as measured by heart rate. | Pre-treatment to post-treatment (10 weeks)
  Change in heart rate to fear generalized from various, perceptually similar stimuli collected during a laboratory fear paradigm. (Discontinued March 2020 due to COVID-19)
Implicit Fear Association Test | Pre-treatment to post-treatment (10 weeks)
  Change in implicit associations for fear-relevant word stimuli
Behavioral Avoidance Test (BAT) | Pre-treatment to post-treatment (10 weeks)
  Change in duration and subjective fear of public speaking in situ
Probability and Cost Questionnaire | Pre-treatment to post-treatment (10 weeks) and follow-up (24 weeks)
  Change in perceived likelihood and perceived consequence of fear-relevant outcomes
Anxiety Sensitivity Index (ASI-3) | Pre-treatment to post-treatment (10 weeks) and follow-up (24 weeks)
  Change in appraisal of harmfulness of symptoms
Positive and Negative Affect Schedule (PANAS 20 item) | Pre-treatment to post-treatment (10 weeks) and follow-up (24 weeks)
  Change in affect
Panic Disorder Severity Scale-Self Report (PDSS-SR) | Weekly throughout the duration of treatment (10 weeks) and once at follow-up (24 weeks)
  Change in panic disorder symptoms
Sheehan Disability Scale (SDS) | Pre-treatment to post-treatment (10 weeks) and follow-up (24 weeks)
  Change in functioning related to mental health
Mini-SPIN | Weekly throughout the duration of treatment (10 weeks) and once at follow-up (24 weeks)
  Change in social anxiety symptoms. Scores on the Mini-SPIN range from 0 to 12 with higher scores indicating higher social anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G Craske, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04048824/Prot_SAP_ICF_000.pdf